CLINICAL TRIAL: NCT00751985
Title: Web-based Ultra-brief Intervention for Heavy Drinkers - a Randomized Controlled Trial Comparing Personalized Normative Feedback With Self-help Material
Brief Title: Web-based Ultra-brief Intervention for Heavy Drinkers Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: National Board of Health, Denmark (Other Government)
Responsible Party: Kit Broholm, National Board of Health Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIPH - 1948b
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2009-05

CONDITIONS: Alcohol Abuse
Keywords: Heavy drinking; Ultra-brief intervention; Brief intervention; Alcohol prevention; Randomized trial; Personal normative feedback; Self-help material; Web-based; Intervention Studies; prevention & control
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Personalized normative feedback (PFI). The PFI was a single-session intervention; it was displayed in a single screenshot and addressed the participant by name. It consisted of a summary of the participant's weekly consumption, a comparison with maximum drinking limits and a graphical comparison of the participant's consumption to the average level in the municipality (gender-specific), followed by information about health and social risks of heavy drinking as well as links for further self-help material and a local alcohol treatment facility.
  Interventions: Other: Personalised normative feedback (PNF)
- 2 (Experimental): Self-help material (SHM). The SHM was a single-session intervention and was displayed in a single screenshot. It consisted of information about maximum drinking limits, followed by information about health and social risks of heavy drinking as well as links for further standardized self-help material and a local alcohol treatment facility.
  Interventions: Other: Self-help material
- 3 (Placebo Comparator): Control
  Interventions: Other: Control

INTERVENTIONS:
Other: Personalised normative feedback (PNF) — The intervention can be classified as a minimal ultra-brief intervention consisting of only a single session.
  The brief personalised normative feedback will comprise the result of the participant's amount of alcohol consumption, previously given in an online questionnaire.
  Alongside, information about alcohol and how it might affect them at their current drinking levels is provided. The feedback is also comparing their drinking, in graphical format, to the average drinking in the municipality concerned. Contact details are also provided about local alcohol treatment possibilities if the participants feel they need further help.
  Arms: 1
Other: Self-help material — The intervention can be classified as a minimal ultra-brief intervention consisting of only a single session.
  The intervention comprises of on-line self-help material informing about the participant's response from an online questionnaire shows that the participant's alcohol consumption exceeds the recommended limits.
  Alongside, information about alcohol and how it might affect them at their current drinking levels is provided. Contact details are also provided about local alcohol treatment possibilities if the participants feel they need further help.
  Arms: 2
Other: Control — The participant is being informed about their allocation to the control group.
  Arms: 3

SUMMARY:
The purpose of the study is to determine whether a web-based ultra-brief intervention, consisting of personalized normative feedback or standardized self-help material, is effective in lowering self reported alcohol use in heavy drinkers.

DETAILED DESCRIPTION:
Background and purpose:

The Danish national board of Health has awarded funds for two studies that will test methods that can be used for effective and early detection of heavy drinkers. The study will be carried out in 12 Danish municipalities in 2008. The study is part of the 'Diet, Smoking, Alcohol and Exercise' nationwide health study of the Danish population. It takes place in 13 municipalities in 2007 and 2008.

The purpose of the study is to determine whether a web-based ultra-brief intervention, consisting of personalized normative feedback or standardized self-help material, is effective in lowering self reported alcohol use in heavy drinkers.

Design:

The experiment is designed as a randomized controlled trial, where heavy drinkers will be allocated to either:

A) an intervention group receiving web-based personalized normative feedback (PFI) B) an intervention group receiving web-based self-help material (SHM) C) a control group receiving nothing.

After 6 and 12 months there will be follow-up and the participants will receive a questionnaire with questions about their alcohol consumption (internetbased and paper).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be invited to the Danish 'Diet, Smoking, Alcohol and Exercise' nationwide health study.
* Participants must have a weekly alcohol consumption above the recommended Danish limits (168 grams of alcohol for women, 252 grams of alcohol for men).

Exclusion Criteria:

* Weekly alcohol consumption less than 168 grams of alcohol for women and 252 grams of alcohol for men.
* Participants who have not informed their email address.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Actual)
Dates: Start 2008-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Reduction of 15% in alcohol consumption with an average volume of approximately 38-41 grams alcohol per week in the PFI group . In the self-help material group we expect that 5 - 10% will reduce their consumption equivalent. | 12 months
  Outcome measure was based on self-reported drinking during a typical week.

CONTACTS AND LOCATIONS:
Overall Officials: Anders B. Gottlieb Hansen, Ph.d.-student, cand.techn.soc, Principal Investigator — University of Southern Denmark, National Institute of Public Health
Locations (1):
- University of Southern Denmark, National Institute of Public Health, Copenhagen, Denmark

REFERENCES:
- [Derived] Hansen AB, Becker U, Nielsen AS, Gronbaek M, Tolstrup JS, Thygesen LC. Internet-based brief personalized feedback intervention in a non-treatment-seeking population of adult heavy drinkers: a randomized controlled trial. J Med Internet Res. 2012 Jul 30;14(4):e98. doi: 10.2196/jmir.1883. PMID 22846542